CLINICAL TRIAL: NCT03706781
Title: A Phase I Study of a Novel Mouthwash Formulation (Cetylpyridinium Chloride 0.05% + Benzydamine HCl 0.15% + Mucus - Adhesive Polymer) Administered Twice a Day for 7 Days to Healthy Subjects in Comparison With Marketed Tantum Verde Bocca Mouthwash Solution
Brief Title: A Novel Mouthwash Formulation CTP/BNZ With Mucus Adhesive Polymer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 030(1C)WO17048
Record Dates: First submitted 2018-04-27; First posted 2018-10-16 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: Phase I; Local tolerability; Systemic Availability; Cetylpyridinium chloride 0.05%; Benzydamine hydrochloride 0.15%; Mucoadhesive polymer; Tantum Verde Bocca
MeSH Terms: interventions — Cetylpyridinium; Benzydamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product CTP/BNZ with mucus adhesive polymer (Experimental): A multiple dose of the Cetylpyridinium Chloride 0.05%+Benzydamine HCl 0.15% (CTP/BNZ) + mucus adhesive polymer is administered to healthy subjects twice a day for 7 days, under fasting conditions in two subsequent periods according to the randomised cross-over design.
  Interventions: Drug: Cetylpyridinium Chloride 0.05% + Benzydamine HCl 0.15% + mucus adhesive polymer
- Reference product CTP/BNZ - Tantum Verde Bocca (Active Comparator): A multiple dose of the Cetylpyridinium Chloride 0.05%+Benzydamine HCl 0.15% (CTP/BNZ) Tantum Verde Bocca is administered to healthy subjects twice a day for 7 days, under fasting conditions in two subsequent periods according to the randomised cross-over design.
  Interventions: Drug: Cetylpyridinium Chloride 0.05% + Benzydamine HCl 0.15%

INTERVENTIONS:
Drug: Cetylpyridinium Chloride 0.05% + Benzydamine HCl 0.15% + mucus adhesive polymer — Test product will be applied twice a day (b.i.d) every 12 h once in the morning and once in the evening for 6 consecutive days (from Day 1 to Day 6) and once in the morning on Day 7 for a total of 13 dose
  Arms: Test product CTP/BNZ with mucus adhesive polymer
Drug: Cetylpyridinium Chloride 0.05% + Benzydamine HCl 0.15% — Reference Product will be applied twice a day (b.i.d) every 12 h once in the morning and once in the evening for 6 consecutive days (from Day 1 to Day 6) and once in the morning on Day 7 for a total of 13 dose
  Other Names: Tantum verde bocca
  Arms: Reference product CTP/BNZ - Tantum Verde Bocca

SUMMARY:
The purpose of the study is to evaluate the local tolerability and the systemic availability of benzydamine, if any, after single and multiple dose treatment with the test formulation containing cetylpyridinium chloride 0.05% + benzydamine hydrochloride 0.15% + mucoadhesive polymer and with the reference formulation Tantum Verde Bocca containing cetylpyridinium chloride 0.05% + benzydamine hydrochloride 0.15% to healthy subjects , under fasting conditions, in two consecutive study periods.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: males/females, 18-55 year old inclusive
3. Body Mass Index: 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the study
6. Contraception and fertility (women only): women of child-bearing potential must be using at least one of the following reliable methods of contraception:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
   2. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner Women of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted.

For all women, pregnancy test result must be negative at screening.

Exclusion Criteria:

1. Electrocardiogram (ECG) 12-leads (supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
5. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study; mouth lesions or any other oral mucosa alteration that may interfere with the aim of the study according to the investigator's opinion
6. Medications: any medications (topical or systemic), including over the counter (OTC) medications, oral rinses and herbal remedies for 2 weeks before the start of the study. Hormonal contraceptives for females will be allowed
7. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
8. Blood donation: blood donations for 3 months before this study
9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2015], caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day)
10. Drug test: positive result at the drug test at screening or Day -1
11. Alcohol test: positive alcohol breath test at Day -1
12. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
13. Pregnancy (females only): positive or missing pregnancy test at screening or Days -1 or 6, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Local Adverse Reactions (ADRs) | Change before and after each administration up to Day 8
  Local ADRs reported by the subjects through a 4-point scale according to a local tolerability scale (degree of severity of reactions from 0 to 3. 0=none; 1=mild 2= moderate; 3= severe) as 0-3 scores for burning sensation, irritation, pruritus, dry mouth, salivary hypersecretion and dysphagia. If the score assigned will be 1, 2 or 3, the local AE will classified as a TEAE of mild, moderate or severe severity, respectively.

SECONDARY OUTCOMES:
Systemic availability of benzydamine (free base) through Cmax. | Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 h after the first dose. Days 7-8: pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 16, 24 h after the last dose.
  Systemic availability of benzydamine (free base) by measurement of plasma concentrations.
Systemic availability of benzydamine (free base) through AUC(0-t). | Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 h after the first dose. Days 7-8: pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 16, 24 h after the last dose.
  Systemic availability of benzydamine (free base) by measurement of area under the plasma concentration-time curve [AUC(0-t)].
Incidence of AEs | Through study completion, an average of three weeks
  General tolerability and safety of the study products assessed through monitoring of AEs including clinically significant abnormalities in laboratory assays (haematology, blood chemistry, urinalysis).
Palatability | Day 7 (after the last dose of each study period).
  Organoleptic properties of the study products evaluated through a ORGANOLEPTIC AND EASE OF USE CHARACTERISTICS questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, Principal Investigator — Cross Research S.A.
Locations (1):
- CROSS Research S.A., Phase I Unit, Via F.A. Giorgioli 14 Phone: Fax: +41.91.63.00.511 Email:, Arzo, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided